CLINICAL TRIAL: NCT00879580
Title: "Prospective Multicenter Observational Study for the Evaluation of the Efficacy of the Cordis Enterprise(TM) Self-expanding Intracranial Stent: Enterprise Stent Aneurysm Treatment (ESAT) Study
Brief Title: Enterprise Stent Aneurysm Treatment (ESAT) Study - France
Acronym: ESAT
Status: Completed | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-FR-001
Record Dates: First submitted 2009-03-31; First posted 2009-04-10 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Intracranial Aneurysm
Keywords: aneurysm; stent; intracranial aneurysm; Ruptured Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-ruptured aneurysms: Patients with intracranial aneurysm(s) requiring an endovascular treatment with a Codman ENTERPRISE stent who have one or more non-ruptured or late ruptured (>30days), intracranial aneurysm.
- Acute ruptured Aneurysms: Patients with intracranial aneurysm(s) requiring an endovascular treatment with a Codman ENTERPRISE stent who have a on or more acute ruptured (<30Days) aneurysms

SUMMARY:
The purpose of this study is to evaluate the morbidity, mortality, and efficacy of use of the Enterprise(TM) stent for the treatment of (ruptured or non-ruptured) intracranial aneurysms.

DETAILED DESCRIPTION:
Per the opinion of the Commission for the Evaluation of Products and Services (CEPP) in France, renewal is contingent upon setup of a prospective morbidity, mortality, and efficacy study. The objective is to follow the stented Subjects for at least 1 year and evaluate the device and practices.

This will be a multicenter study involving up to 15 interventional neuroradiologists in France. Subjects presenting with ruptured or non-ruptured aneurysms for whom simple or balloon assisted endovascular treatment is considered impossible or insufficient by the interventional neuroradiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with one or more CODMAN ENTERPRISE™ stents and who present one or more ruptured or non-ruptured intracranial aneurysms assessed by angiography
* Agreement to take part in the study by the patient, or a representative of the patient in case of patient inability, after being informed by the investigator and have received information letter.

Exclusion Criteria:

* Minors <18 years of age
* Patient implanted for the same aneurysm with a CODMAN ENTERPRISE™ stent in association with one or more stents from a different brand.
* Patient who does not accept to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with ruptured or non-ruptured aneurysms for whom simple or balloon-assisted endovascular treatment is considered impossible or insufficient by the interventional neuroradiologist.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Morbidity and Mortality | Day 30 and 1 year post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Megerian, MD, PhD, Study Director — Codman & Shurtleff
Locations (14):
- France (14):
  - CHU Amiens, Amiens
  - Jean Minjoz Hospital, Besançon
  - Pellegrin Hospital, Bordeaux
  - Albert Michallon Hospital, Grenoble
  - Roger Salengro Hospital, Lille
  - Timone Hospital, Marseille
  - Lariboisiere Hospital, Paris
  - La Pitie Salpetiere Hospital, Paris
  - Pitie Salpetriere Hospital, Paris
  - La Pitie Salpetriere Hospital, Paris
  - Rothschild Foundation, Paris
  - Beaujon Hospital, Paris
  - White House Hospital, Reims
  - Purpan Hospital, Toulouse